CLINICAL TRIAL: NCT04139343
Title: The Role of Motor Unit Number Estimation (MUNE) in Adults With Spinal Muscular Atrophy (SMA)
Brief Title: Motor Unit Number Estimation (MUNE) in Adults With Spinal Muscular Atrophy (SMA)
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Cure SMA (Other)
Responsible Party: Principal Investigator, Bakri Elsheikh, Professor, Ohio State University
Other Study IDs: 2006H0207
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Spinal Muscular Atrophy
Keywords: nusinersen; Spinraza; MUNE; CMAP
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- SMA cohort: Individuals who have a diagnosis of SMA who are NOT receiving Spinraza (nusinersen).
- SMA Spinraza cohort: Individuals who have a diagnosis of SMA who are receiving Spinraza (nusinersen).
- Control cohort: Control participants will only come to a baseline visit and the only tests that will be completed are the EMG Measures (MUNE, CMAP, decomposition EMG) and EIM. There will be no further testing for those participants. This visit will take approximately 30-60 minutes. A total of 40 control participants are being recruited for this study.

SUMMARY:
The primary objective of this research protocol is to study and follow the course of motor neuron loss in individuals with spinal muscular atrophy (SMA) using the electrophysiological technique of motor unit number estimation (MUNE). This study is based on the hypothesis that the electrophysiological technique of motor unit number estimation (MUNE) and compound muscle action potential (CMAP) provide sensitive indicators to assess the severity and progression of disease in adults with SMA.

DETAILED DESCRIPTION:
This is a prospective pilot study to determine MUNE and CMAP values in a population of adults with SMA, assess how these electrophysiologic parameters change over time, and explore how well these parameters correlates with other outcome measures in SMA, including functional scales (SMAFRS and SF-36) and muscle strength (by MMT, MVICT, 6 minute walk test, time to climb 4 stairs and handheld myometry). The study was started in 2006 with 4 visits. It was initially intended to measure baseline and variability of values at baseline, 6 months, 10-14 months, and 20-24 months to better characterize the disease and to validate measurements as suitable outcome measures to be used in future therapeutic trials on adults. Individuals who do not take nusinersen would continue on this visit plan.

With the addition of the FDA approved drug nusinersen for SMA we would like to follow people who are receiving that treatment more frequently. The visits will fall in relationship to their treatment doses. Those patients who are receiving nusinersen will come in at a baseline visit that will be1 to 6 weeks prior to first treatment. Then they would follow-up one to 2.5 weeks after each treatment dosing that happens quarterly after the initial loading dose. There will be 10 visits over 3 years. The visits will occur at baseline, 2, 6, 10, 14, 18, 22, 26, 30, and 34 months. These additional visits will allow for better uniform monitoring of the response to treatment and resubmission to insurance providers. Additional long term data will be collected from interested/available patients every 2-3 years up to a max of fifteen years. Being followed long term would add 4-6 visits over 12 years. If subjects completed the study course in the past and are now starting nusinersen (SPINRAZA), those individuals are able to enroll again.

A total of 100 people with SMA will be enrolled in this trial. This will allow for two cohorts of people with SMA; those receiving treatment and those not receiving treatment.

Control participants will only come to a baseline visit and the only tests that will be completed are the EMG Measures (MUNE, CMAP, decomposition EMG) and EIM. There will be no further testing for those participants. This visit will take approximately 30-60 minutes. A total of 40 control participants are being recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults age 17 to 70 with SMA type 2 or 3. The diagnosis of SMA must be documented by the homozygous deletion of both SMN1 genes on standard genetic tests for the disorder, and the determination of type 2 SMA by history of ability to maintain a sitting position when placed, or type 3 by the ability to stand and walk independently. Wheelchair mobile patients will not be excluded from the study.

  2. Interest in participating and the ability to travel to the study site on an agreed upon date on four occasions over a total interval of twenty-four months.

  3. Be in good health with the exception of SMA. Assessments will be rescheduled for a later date in the event of any intercurrent illness that might affect performance on the assessment.

Inclusion criteria for control subjects:

1. Healthy adults age 17 to 70
2. Interest in participating and the ability to travel to the study site

Exclusion Criteria:

- Patients unable to tolerate the assessment by virtue of associated medical conditions, respiratory failure with ventilator dependence, or an obligatory need for orthotics that cannot be removed during the evaluation.

2. Patients who are, in the investigator's opinion, mentally or legally incapacitated, preventing informed consent, or is unable to read and understand written material including the consent 3. Patients with a pacemaker or cardiac device

Exclusion criteria for control subjects:

1. Subjects with any neurological disorder
2. Subjects with chronic medical illness that will interfere with their ability to tolerate the study
3. Subjects who are, in the investigator's opinion, mentally or legally incapacitated, preventing informed consent, or is unable to read and understand written material including the consent.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals between 17-70 years of age who have been diagnosed with spinal muscular atrophy (SMA) regardless of current medical intervention (e.g., Spinraza).
  The control group will consist primarily of (but not restricted to) family members of those enrolled in the study who have a diagnosis of SMA.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MUNE | up to 15 years
  The primary objective of this proposal is to study and follow the course of motor neuron loss in adults with spinal muscular atrophy (SMA) using the electrophysiological technique of motor unit number estimation (MUNE). This study is based on the hypothesis that the electrophysiological technique of motor unit number estimation (MUNE) can provide sensitive indicator data to assess the severity and progression of disease in adults with SMA.
CMAP | up to 15 years
  The primary objective of this proposal is to study and follow the course of motor neuron loss in adults with spinal muscular atrophy (SMA) using the electrophysiological technique of compound muscle action potential (CMAP). This study is based on the hypothesis that the electrophysiological technique of compound muscle action potential (CMAP) can provide sensitive indicator data to assess the severity and progression of disease in adults with SMA.

SECONDARY OUTCOMES:
EIM | up to 15 years
  Secondary Objective is to see if electrical impedance myography (EIM) correlates to the electrophysiological testing (see Primary Outcome measures: MUNE and CMAP).
Nusinersen | up to 15 years
  Explore the changes in outcome measures in patients treated with nusinersen
Treatment insurance approval and safety | up to 15 years
  Explore the insurance approval process, patient acceptance, and side effects of the newly approved FDA treatment of nusinersen.

CONTACTS AND LOCATIONS:
Overall Officials: Bakri Elsheikh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided